CLINICAL TRIAL: NCT00791193
Title: Pharmacokinetic Evaluation of the Relative Bioavailability of Three Paliperidone Extended Release (ER) Formulations With Different in Vitro Release Profiles, and Comparison to Paliperidone Immediate Release (IR), in Healthy Male Subjects
Brief Title: A Pharmacokinetic Study of the Relative Bioavailability of Paliperidone ER Formulations With Different Release Profiles and a Comparison to Paliperidone IR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR013474
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2010-04

CONDITIONS: Schizophrenia
Keywords: Paliperidone ER; Antipsychotic drugs; Schizophrenia; Mood disorders
MeSH Terms: conditions — Schizophrenia; Mood Disorders | interventions — Paliperidone Palmitate

INTERVENTIONS:
Drug: Paliperidone ER

SUMMARY:
The primary purpose of this study is to evaluate the pharmacokinetics and relative bioavailability of paliperidone ER formulations with slow, target, and fast in vitro release rates after administration of a single 12 mg dose. The slow and fast releasing ER tablets have in vitro release rates outside the current commercial specifications. Therefore, in order to support widening of the specification limits, this study will be performed. The target formulation to be used is representative of the commercial formulation. Other objectives of this study are 1) to compare the relative bioavailability of paliperidone ER formulations with slow, target, and fast in vitro release rates to the paliperidone IR formulation; 2) to explore the in vitro in vivo correlation (IVIVC) for the paliperidone ER formulation; and 3) to evaluate the safety and tolerability of the different paliperidone ER formulations.

DETAILED DESCRIPTION:
This is a randomized, open-label, 4-way crossover, single dose study in healthy male volunteers to evaluate the pharmacokinetic profiles of paliperidone ER tablets with slow, target, and fast in vitro release rates and paliperidone IR. The study consists of a 21 day screening phase, an open-label treatment phase consisting of 4 single-dose treatment periods (IR, slow, fast, and target formulations), and an end-of-study or early withdrawal phase. A 10- to 21 day washout period (i.e., >5 times the half-life) will separate each study drug administration (i.e., each open label treatment period). In the first period, all volunteers are given a 1-mg dose of paliperidone IR solution, administered as a single oral dose under fasted conditions (Treatment A). On Day 1 of Period 2, prior to study drug administration, all volunteers will be randomly assigned to 1 of 6 possible treatment sequences to ensure that they receive all of the following treatments, one in each period: 12-mg paliperidone ER tablet with a target in vitro release under fasted condition (Treatment B); 12-mg paliperidone ER tablet with a slow in vitro release under fasted condition (Treatment C); 12-mg paliperidone ER tablet with a fast in vitro release under fasted condition (Treatment D). In each treatment period, volunteers will enter the study center at least 10 hours before the study drug administration on Day 1 and will remain there until after collection of the 96 hour pharmacokinetic samples on Day 5 if the investigator considers that the volunteer is ready for discharge. It is expected that the differences in the in vitro release rate will not affect the relative bioavailability of paliperidone in vivo. Safety and tolerability of the different paliperidone ER formulations will be monitored throughout the study.

Single oral doses of paliperidone ER 12 mg tablets with different release rates (target, fast, and slow); single oral dose of paliperidone IR 1 mg

ELIGIBILITY:
Inclusion Criteria:

* Must agree to use an efficient method of birth control as deemed appropriate by the investigator and to not donate sperm during the study and for 3 months after receiving the last dose of study drug
* Body mass index (weight [kg]/height [m2]) between 18 and 30 kg/m2 (inclusive), and body weight not less than 50 kg
* Blood pressure (after the volunteer is supine for 5 minutes) between 100 and 140 mmHg systolic, inclusive, and between 50 and 90 mmHg diastolic. Pulse rate measured over 60 seconds should be between 40 and 100 beats per minute (bpm)
* Non-smoker

Exclusion Criteria:

* History of or current significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the volunteer
* History or presence of circumstances that may increase the risk of the occurrence of torsade de pointes and/or sudden death in association with the use of drugs that prolong the QTc interval, including: bradycardia (heart rate < 40 bpm on the ECG), clinically significant abnormality on the ECG, demonstration of repeated prolonged QTcF > 450 ms (QTc interval corrected for heart rate using Fridericia's formula), as measured on more than one ECG (either during screening, or from prior medical record)
* The following cardiac conditions: sick sinus syndrome, complete AV block, congestive heart failure, polymorphic ventricular tachycardia
* Clinically relevant hypocalcemia, hypokalemia or hypomagnesemia
* Presence of congenital prolongation of the QT interval (Romano-Ward Syndrome, Jervell and Lange-Nielsen syndrome)
* History of any cancer, with the exception of basal cell carcinoma: Clinically significant abnormal values for hematology, clinical chemistry or urinalysis at screening or at admission to the study center, in the opinion of the investigator
* Clinically significant abnormality on physical examination, in the opinion of the investigator
* At screening, has signs of orthostatic hypotension defined as a decrease in systolic ( > 20 mmHg) or diastolic (> 10 mmHg) blood pressure after standing for at least 2 minutes, that is associated with an increase in pulse rate of >15 bpm compared with supine measurements
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for paracetamol (acetaminophen) or ibuprofen, within 14 days before the first dose of the study drug is scheduled

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2007-03; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetics and relative bioavailability of paliperidone ER formulations with different in vitro release rates (slow, fast) compared to the target formulation after a single 12 mg dose.

SECONDARY OUTCOMES:
To evaluate the relative bioavailability of paliperidone ER formulations with different in vitro release rates compared to the paliperidone IR formulation, to explore an IVIVC for the paliperidone ER formulation, and to assess safey and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A pharmacokinetic study of the relative bioavailability of paliperidone ER formulations with different release profiles and a comparison to paliperidone IR — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=761&filename=CR013474_CSR.pdf